CLINICAL TRIAL: NCT05473481
Title: Dynamic EchoCardiographic Optimisation REsponse Study (Studio Sulla Risposta All'Ottimizzazione Dinamica Ecocardiografica)
Brief Title: Dynamic EchoCardiographic Optimisation REsponse Study
Acronym: DECORE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Massimo Saviano, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 2752/6065
Record Dates: First submitted 2022-07-19; First posted 2022-07-26 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the effects of heart rate optimization and guided A-V and V-V delay from color Doppler echocardiography, in subjects affected by heart failure with reduced ejection fraction and CRT-D device wearers who did not respond to device implantation in clinical, electrophysiological, and other terms.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be 18 to 85 years of age inclusive, at the time of signing the informed consent form;
2. Heart failure with ventricular ejection fraction left <45%;
3. Presence of CRT-D devices in a non-responder patient for cardiac resynchronization
4. NYHA >II;
5. Resting heart rate <65 beats per minute;
6. Biventricular pacing >97%.

Exclusion Criteria:

1. Age <18 and >85 years;
2. Insufficient functional capacity to complete the tests required by the research protocol;
3. Permanent Atrial Fibrillation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects affected by heart failure with reduced ejection fraction and CRT-D device wearers, who did not respond to the implantation of the device in clinical and electrophysiological terms.
Sampling Method: Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of acute heart failure episodes | Baseline to 12 months post discharge
  Number of worsening HF episodes requiring hospitalization
Change in left ventricular ejection fraction (LVEF) | Baseline to 12 months post discharge
  An echocardiogram will be performed at specific study visits and LEVF will be measured
Echocardiofic changes of diastolic left ventricular function | Baseline to 12 months post discharge
  An echocardiogram will be performed at specific study visits and LVESV and LVEDV will be

SECONDARY OUTCOMES:
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline to 12 months post discharge
  This is a disease-specific health status instrument composed of 23 items that quantify the domains of physical limitation, symptoms, self-efficacy, social limitation, and quality of life limitation due to HF. Scores range from 0 to 100. For the KCCQ overall summary score, a small but clinically meaningful change is ≥ 5 points.
Change in NYHA class | Baseline to 12 months post discharge
  Measures of New York Heart Association functional class stratified I to IV at baseline and at each scheduled time.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Maggiore Policlinico di Milano, Milan, MI, Italy